CLINICAL TRIAL: NCT01312727
Title: Phenotypical and Genetic Characterization of Adult Hereditary Chronic Tubulointerstitial Renal Diseases
Brief Title: Hereditary Tubulointerstitial Nephritis
Acronym: NTIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: P081258
Record Dates: First submitted 2011-02-22; First posted 2011-03-11 (Estimated); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Nephritis, Interstitial; Chronic Renal Failure; Gout; Renal Cysts
Keywords: Tubulointerstitial renal diseases; Hereditary renal diseases; Uromodulin; Renin gene
MeSH Terms: conditions — Nephritis, Interstitial; Kidney Failure, Chronic; Gout | interventions — Blood Specimen Collection; Phenotype; Genotype

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HTIN (Other): HTIN
  Interventions: Other: Blood and urine sample collections

INTERVENTIONS:
Other: Blood and urine sample collections — phenotype and genotype analysis, biological analysis
  Other Names: phenotype and genotype analysis, biological analysis

SUMMARY:
The aim of this study is to identify families with hereditary chronic tubulointerstitial renal diseases , characterize the phenotype and screen for mutations in known genesis (UMOD, REN, TCF2, NPHP1). Genome wide analysis will be performed in families without mutations identified.

DETAILED DESCRIPTION:
* Inclusion of affected subjects with familial history of chronic renal failure, early gout ,renal cysts in several hospital in France
* Characterization of the phenotype; dosage of the urinary uromodulin in all subjects
* Collect DNA samples
* Screen for UMO mutations first
* Then for REN or TCF2 depending on the phenotype
* Validate the use of the dosage of urinary uromodulin for the diagnosis of UMOD associated disease.
* Identify new genes responsible for hereditary HTIN (Hereditary Tubulointerstitial Nephritis).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* HTIN of unknown cause
* Chronic renal failure defined by a eGFR (estimated Glomerular Filtration Rate) estimated according to MDRD (Modification of the Diet in Renal Disease) < 60ml / min / 1,73m2.
* At least two siblings affected by gout before 40 years or by chronic renal failure.
* Affiliated or benefiting from a national insurance
* Signature of the enlightened consent.

Exclusion Criteria:

* Endstage renal failure before the age of 18 years in all affected subjects of the family.
* Microscopic or macroscopic persistent hematuria, or proteinuria > 1gramme / 24hours.
* Other potential cause of TIN (Tubulointerstitial Nephritis): pyelonephritis, drug toxicity.
* High blood pressure known for more than 10 years before the discovery of the renal disease.
* Major cardiovascular before the discovery of the renal disease.
* Chronic auto-immune or infectious disease.
* Polycystic kidney disease with increased of the size of the kidneys

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2010-11; Primary Completion 2014-02 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Genotype of HTIN | after 18 months
  Number of patients/families with mutations in known genes responsible for HTIN

SECONDARY OUTCOMES:
Uromodulin dosage in urine | at 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Knebelmann, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker Enfants Malades, Paris, France

REFERENCES:
- [Result] Saei H, Moriniere V, Heidet L, Gribouval O, Lebbah S, Tores F, Mautret-Godefroy M, Knebelmann B, Burtey S, Vuiblet V, Antignac C, Nitschke P, Dorval G. VNtyper enables accurate alignment-free genotyping of MUC1 coding VNTR using short-read sequencing data in autosomal dominant tubulointerstitial kidney disease. iScience. 2023 Jun 17;26(7):107171. doi: 10.1016/j.isci.2023.107171. eCollection 2023 Jul 21. PMID 37456840